CLINICAL TRIAL: NCT01612182
Title: The Incidence of Extended-spectrum β-lactamase (ESBL) Klebsiella Pneumonia in Patient on Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Hoseok Koo, Nephrology division, Department of Internal Medicine, Inje University
Other Study IDs: ESBL 2012-1
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: End-stage Renal Disease
Keywords: end-stage renal disease; renal replacement therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Replacement Therapy

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- ESBL(+) Klebsiella pneumonia: All the patient who's the culture result showed ESBL(+) Klebsiella pneumonia in any site during hospitalization
  Interventions: Other: renal replacement therapy
- ESBL(-) Klebsiella pneumonia: All the patient who's the culture result showed ESBL(-) Klebsiella pneumonia in any site during hospitalization
  Interventions: Other: renal replacement therapy

INTERVENTIONS:
Other: renal replacement therapy — renal replacement therapy : hemodialysis and/or CRRT(continuous renal replacement therapy )

SUMMARY:
The prevalence of ESBL Klebsiella pneumonia was higher in patient with renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* The age of patient was between 18 yrs and 79 yrs.
* The patient who showed Klebsiella pneumonia in 1st culture result of any site during hospitalization

Exclusion Criteria:

* The level of serum albumin was below 2.0 or over 5.0
* The level of AST or ALT was 2 times of normal level or the level of bilirubin was over 2.0 mg/dL during 1month.
* The level of Body mass index was below 15 or over 30
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients had admitted in single center
Sampling Method: Non-Probability Sample
Enrollment: 1289 (Actual)
Dates: Start 2012-03; Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The prevalence of ESBL Klebsiella pneumonia in renal replacement therapy | During hospitalization
  The prevalence of ESBL Klebsiella pneumonia in renal replacement therapy during hospitalization up to 8 years (from 2004 to 2011)

SECONDARY OUTCOMES:
The prevalence of ESBL Klebsiella pneumonia in patient with pneumonia and renal replacement therapy | during hospitalization
  The prevalence of ESBL Klebsiella pneumoina in patient with pneumonia and renal replacement therapy during hospitalization up to 8 years (from 2004 to 2011)

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Seoul Paik hospital Instituional Board Review, Seoul, Je Dong 2ga, Jung Gu, South Korea